#### Cover page - statistical analysis plan

#### Title

Obstetric outcome in pregnancies treated with laparoscopic cerclage: an observational study in a Danish cohort

## **Roles and Responsibility**

Study group

Principal investigator; Lise Qvirin Krogh, MD<sup>1</sup>

Daily supervisor; Julie Glavind, PhD, Associate Professor, Consultant in Obstetrics<sup>1</sup>

Study Sponsor & co-investigator; Niels Uldbjerg, Professor in Obstetrics<sup>1</sup>

Co-investigator; Iben Sundtoft, PhD, Associate Professor, Consultant in Obstetrics<sup>2</sup>

Co-investigator; Lea Kirstine Hansen, MD<sup>1</sup>

Co-investigator; Rikke Bek Helmig, Consultant in Obstetrics<sup>1</sup>

Co-investigator; Axel Forman, Professor Emeritus in Gynecology<sup>1</sup>

#### **Conflicts of interest**

The members of the study group have no conflicts of interest to declare. The study sponsor has no ultimate authority over any aspects of the study design, conduct, or reporting.

## **Trial registration**

The study is registered at clinicaltrials.gov using the administrative authorities of Aarhus University (UAarhus). NCT05863481.

#### **Funding**

Funding for the study is provided as a part of a larger grant by the Novo Nordic Foundation.

<sup>&</sup>lt;sup>1</sup>Department of Obstetrics and Gynecology, Aarhus University Hospital, Denmark

<sup>&</sup>lt;sup>2</sup>Department of Obstetrics and Gynecology, Regional Hospital Gødstrup, Denmark

## Statistical analysis plan

Statistics will be descriptive and data will be presented with counts and percentages for categorical variables, mean and standard deviation for continuous Gaussian distributed variables, and median and interquartile range for continuous non-Gaussian variables. Proportions will be presented with a 95% confidence interval for the dichotomous outcomes.

Subgroup analyses of the primary outcome will be undertaken for the following subgroups:

- Prior versus no prior cesarean delivery at time of laparoscopic cerclage
- Prior versus no prior conisation at time of laparoscopic cerclage
- Placement of laparoscopic abdominal cerclage before or during early pregnancy

STATA will be used for data management and analyses.

Examples of anticipated tables is shown below.

**Table 1.** Maternal Characteristics upon laparoscopic cerclage placement

| 1 | n |
|---|---|
| Age, years | mean (range) |
| Smoking | no. (%) |
| Body Mass Index (kg/m²) | median (interquartile range) |
| Parity | median (interquartile range) |
| Previous conization | no. (%) |
| 0 | no. (%) |
| 1 conus | |
| 2+ | |
| Previous caesarean delivery Performed as emergency caesarean | no. (%) |
| - , | no. (%) |
| Previous uterine surgery | • • |
| Placement of laparoscopic ceclage during pregnancy | no. (%) |
| ndications for the laparoscopic cerclage placement | |
| <ul> <li>a) Previous emergency/laboring cesarean delivery followed by a spontaneous<br/>singleton late miscarriage or preterm birth from 16+0 to 28+0 weeks</li> </ul> | no. (%) |
| <ul> <li>Previous elective vaginal cerclage placement but nonetheless a spontaneou<br/>late miscarriage or preterm birth between 14+0 and 28+0 weeks (= failed<br/>vaginal cerclage)</li> </ul> | no. (%) |
| <ul> <li>Previous ultrasonography-indicated emergency cerclage with preterm birth<br/>between 14+0 and 28+0 weeks</li> </ul> | no. (%) |
| d) Conization and a short pre-pregnancy cervix | no. (%) |
| <ul> <li>e) Two or more deliveries in gestational age 16+0 to 28+0 weeks and a clinical<br/>diagnosis of cervical insufficiency</li> </ul> | no. (%) |
| f) Three or more deliveries in gestational age 16+0 to 36+6 weeks | no. (%) |
| g) Others | no. (%) |

Table 2. Characteristics laparoscopic cerclage procedure

| n | n |
|---|---|
| Additional procedures performed during surgery | no. (%) |
| Performed in Day Surgery | no. (%) |
| Year of surgery | |
| 2011 trough 2014 | no. (%) |
| 2015 trough 2018 | no. (%) |
| 2019 trough 2022 | no. (%) |
| Early complications | |
| Conversion to laparotomy during surgery | no. (%) |
| Haemorrhage > 500 ml | no. (%) |
| Postoperative infection treated at hospital | no. (%) |
| Damage to internal organs | no. (%) |
| Need for re-operation | no. (%) |
| Admission to Intensive Care Unit | no. (%) |
| Thromboembolic events | no. (%) |
| Maternal cardiopulmonary arrest | no. (%) |
| Maternal death | no. (%) |
| Late complications | |
| Erosion into the vagina treated in hospital | no. (%) |
| Pain complaints from the stiches leading to intervention in pregnancy | no. (%) |
| Other complications from the cerclage leading to intervention in hospital | no. (%) |

Table 3. Pregnancy outcomes and neonatal survival subsequent to laparoscopic cerclage placement

| Pregnancy | n | Neonatal | Neonatal | | | Time of n | niscarriages | or delivery | | Gestational |
|---|---|---|---|---|---|---|---|---|---|---|
| no. | | survival | survival<br>without major<br>morbidity | ≤16 GW | ≤22 GW | ≤28 GW | ≤32 GW | ≤34 GW | ≤37 GW | age |
| 1 | n | prop. (95% CI) | prop. (95% CI) | no. (%) | no. (%) | no. (%) | no. (%) | no. (%) | no. (%) | median (IQR) |
| 2 | n | prop. (95% CI) | prop. (95% CI) | no. (%) | no. (%) | no. (%) | no. (%) | no. (%) | no. (%) | median (IQR) |
| 3 | n | prop. (95% CI) | prop. (95% CI) | no. (%) | no. (%) | no. (%) | no. (%) | no. (%) | no. (%) | median (IQR) |
| 4 | n | prop. (95% CI) | prop. (95% CI) | no. (%) | no. (%) | no. (%) | no. (%) | no. (%) | no. (%) | median (IQR) |
| 5 | n | prop. (95% CI) | prop. (95% CI) | no. (%) | no. (%) | no. (%) | no. (%) | no. (%) | no. (%) | median (IQR) |

| Obstetric outcome in pregnancie | s treated with laparoscopic cerclage |
|---------------------------------|---------------------------------------|
| | Statistical analysis plan version 1.0 |

| Table 4 Time intermed | Obstetric outcome in pregnancies treated with Japard |
|---|---|
| <b>Table 4.</b> Time intervals | Statistical analysis i |

median (IQR) Time from the laparoscopic cerclage to first pregnancy (years and days)

# **Table 5.** Characteristics of live born neonates

| n | n |
|--------------------------|--------------|
| Gestational age at birth | no. (%) |
| Birth weight (g) | median (IQR) |